CLINICAL TRIAL: NCT03999866
Title: Awake Airway Assessment With Video Laryngoscopes
Brief Title: Preoperative Assessment of Difficult Laryngoscopy Using Different Videolaryngoscopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Diagnostic
Other Study IDs: KİA 2019/18
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Assessment; Difficult Airway Intubation; Preoperative
Keywords: airtraq; c-mac; d-blade; mcgarth mac x-blade; prediction; difficult airway

STUDY DESIGN:
Intervention Model Description: We used these 4 video laryngoscopes ( c-mac, d-blade, macgrath mac x-blade and airtraq) on the same patient.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- satisfaction of instructor (Active Comparator): visual analogy scale of the satisfaction of the instructor was recorded
  Interventions: Device: airtraq; Device: mcgrath mac x-blade; Device: storz c-mac; Device: storz d-blade
- satisfaction of the patient (Active Comparator): visual analogy scale of the satisfaction of the patient was recorded
  Interventions: Device: airtraq; Device: mcgrath mac x-blade; Device: storz c-mac; Device: storz d-blade
- duration of view (Active Comparator): duration of the visualization the vocal cords was recorded
  Interventions: Device: airtraq; Device: mcgrath mac x-blade; Device: storz c-mac; Device: storz d-blade

INTERVENTIONS:
Device: airtraq — airtraq videolaryngoscope
  Other Names: videolaryngoscope
Device: mcgrath mac x-blade — mcgarth mac videolaryngoscope
  Other Names: videolaryngoscope
Device: storz c-mac — storz c-mac videolaryngoscope
  Other Names: videolaryngoscope
Device: storz d-blade — storz d-blade video laryngoscope
  Other Names: videolaryngoscope

SUMMARY:
preoperative assessment of difficult airways are the subject of debate. Now, measuring the thyromental distance or evaluating the mallampati score, mandible protrusion or body mass index still not 100% specifically say anything. We compare 4 different video laryngoscopes for preoperative assessment of difficult laryngoscopy.

DETAILED DESCRIPTION:
preoperative assessment of difficult airways are the subject of debate. Now, measuring the thyromental distance or evaluating the mallampati score, mandible protrusion or body mass index still not 100% specifically say anything. all patients were pre oxygenated with 100% oxygen with nasal canulla during the whole procedure. We administered 0.07 mgr/kg remifentanil for minimum 3 minutes and continue this infusion during the procedure. The patients airway topicalized by 10% lidocaine spray. We enroll 20 patients undergoing elective surgery.

We compare 4 different video laryngoscopes for preoperative assessment of difficult laryngoscopy in the same patient. We evaluate the patient and the instructors satisfaction with the visual analogy scale and the visualization time. Demographic vary,ables and the airway characteristics of patients. We assess the cormack lehane view of these videolaryngoscopes with or without cricoid pressure. and the occurrence of gag reflex as well.

ELIGIBILITY:
Inclusion Criteria:- > 18 years or <60 years of age,

* body mass index < 30
* no difficult airway history or predictor,
* no respiratory tract infections for ten days,

Exclusion Criteria: BMI > 35, < 18 or > 60 years of age, expected difficult airway, pregnant

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
satisfaction of the instructor: visual analogy scale | 2 minutes
  visual analogy scale of the satisfaction

SECONDARY OUTCOMES:
satisfaction of the patient: visual analogy scale | 2 minutes
  visual analogy scale of the satisfaction
duration view | 10 seconds
  time frame from the device enter the oral cavity till the vocal cords visualized

CONTACTS AND LOCATIONS:
Overall Officials: Zehra I Arslan, Study Chair — Associate Professor
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No